CLINICAL TRIAL: NCT00381381
Title: A Multi-center Study for the Clinical Response of Choline Acetyltransferase and Apolipoprotein Epsilon Gene Polymorphisms to Donepezil in Alzheimer's Disease
Brief Title: The Clinical Response of Choline Acetyltransferase and Apolipoprotein Epsilon Gene Polymorphisms to Donepezil in Alzheimer's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EKI-6-004
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Results first posted 2012-07-27 (Estimated); Last update posted 2022-01-04 (Actual); Status verified 2010-07

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Donepezil — 2.5mg once daily for the first 7 days, 5mg once daily for the next 3 weeks, after then the dose can be increased 10mg once daily under the investigator's decision.
  Other Names: Aricept

SUMMARY:
This study attempts to differentiate the clinical responses of Choline Acetyltransferase and Apolipoprotein Epsilon gene polymorphism to donepezil in Alzheimer's Disease patients.

ELIGIBILITY:
Inclusion criteria:

1. Age: 60 - 90 years old.
2. CDR: 0.5 - 2.0.
3. Patients who do not have severe depressive symptoms that affect cognition on depression scale of CERAD-K(C), GDS-K: 19 and below.
4. Modified Hachinski Ischemic Score (Rosen, et. al., 1979): 3 and below.
5. NINCDS-ADRDA criteria: Probable AD.

Exclusion criteria:

1. Patients who have delusions and other conscious dysfunction.
2. Patients who have neurologic diseases such as Parkinson's disease, stroke, tumor, normal pressure hydrocephalus, etc., on history and neurologic examination.
3. Patients who have history of infectious and inflammatory brain disease owing to virus, fungus and syphilis.
4. Patients with severe cerebrovascular pathology.
5. Patients who have present history of major psychological diseases such as depression and mania according to DSM-IV criteria.
6. Patients who have history of alcoholism or drug addiction.
7. Patients who have severe depressive symptoms that affect cognition on depression scale of CERAD-K.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2006-05-31 (Actual); Primary Completion 2008-08-31 (Actual); Study Completion 2008-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jihee Mun, Study Director — Eisai Korea Inc.
Locations (15):
- South Korea (15):
  - Seoul National University Bundang Hospital, Bundang
  - Hallym University Medical Center, Changwon
  - Kangwon National University Hospital, Chuncheon
  - Kunkuk University Chungju Hospital, Chungju
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Gyeonggi Province Geriatric Hospital, Gyeonggi-do
  - Uijeongbu St. Mary's Hospital, Gyeonggi-do
  - Jeju National University Hospital, Jeju City
  - Jeonju City Welfare Hospital, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Inje University Pusan Paik Hospital, Pusan
  - Kunkuk University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 15 centers in Korea during the period of June 2006 to August 2008.
Groups:
- Donepezil: Initial dose was 2.5 mg/day, and the maximum dose was 10 mg/day.
Period: Overall Study
Arm/Group | Donepezil
Started | 199
Completed | 135
Not Completed | 64
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 52
Not completed — Withdrawal by Subject | 9

BASELINE CHARACTERISTICS:
Arm/Group | Donepezil
Number analyzed (Participants) | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.6 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136
  Male | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 199
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: CERAD-K (the Korean Version of the Consortium to Establish a Registry for Alzheimer's Disease)
Description: CERAD-K includes: Verbal Fluency-number of kinds of animal patients listed per minute, ranges from 0, no maximum point fixed.Boston Naming Test is naming objects (0-15). Mini-Mental State Examination in the Korean version of CERAD Assessment Packet (0-30). Word List Memory (0-30). Construction Praxis is from 0-11. Word List Recall and Word List Recognition ranges from 0-10.Construction Recall (0-11).
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Donepezil
Number analyzed (Participants) | 135
Units on Scale
  Verbal Fluency | 8.28 (3.71)
  Boston Naming Test | 7.31 (3.25)
  MMSE-KC | 17.86 (5.25)
  Word List Memory | 10.62 (6.20)
  Construction Praxis | 7.61 (2.71)
  Word List Recall | 1.98 (1.99)
  Word List Recognition | 4.64 (3.24)
  Construction Recall | 2.11 (2.71)

2. Secondary Outcome: Neuropsychiatry Inventory (NPI)
Description: NPI score after treatment. NPI includes 12 sections which are Delusions, Hallucinations, Agitation, Depression, Anxiety, Euphoria, Apathy, Disinhibition, Irritability, Aberrant motor behavior, Night-time behaviors and Appetite and eating disorders. The score of each section ranges from 0 to 12, and higher score means higher severity and frequency of the neuropsychiatric disturbances.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Donepezil
Number analyzed (Participants) | 135
Units on Scale
  Delusions | 0.49 (1.85)
  Hallucinations | 0.12 (0.69)
  Agitation | 0.54 (1.56)
  Depression | 0.76 (1.82)
  Anxiety | 0.70 (2.10)
  Euphoria | 0.02 (0.19)
  Apathy | 1.44 (2.69)
  Disinhibition | 0.28 (1.19)
  Irritability | 0.67 (1.93)
  Aberrant motor behavior | 0.44 (1.71)
  Night-time behaviors | 0.40 (1.68)
  Appetite and eating disorders | 0.43 (1.46)

3. Secondary Outcome: GDS-K (Geriatric Depression Scale-Korean) Score After Treatment
Description: GDS-K score after treatment. Geriatric Depression Scale is a basic screening measure for depression in older adults. It ranges from 0 to 30, and higher score represents more depressed.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Donepezil
Number analyzed (Participants) | 135
Units on Scale | 11.69 (6.42)

4. Primary Outcome: CERAD-K
Description: CERAD-K includes: Trail making test A and B is scored by the time spent to link randomly arranged numbers and alphabets in correct order. Except Trail making test A and B, higher score presents better condition.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: Second
Arm/Group | Donepezil
Number analyzed (Participants) | 135
Second
  Trail making test A | 206.64 (126.94)
  Trail making test B | 290.88 (30.20)

ADVERSE EVENTS:
Arm/Group | Donepezil
Serious Adverse Events (participants affected / at risk) | 4/199
Other Adverse Events (participants affected / at risk) | 30/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donepezil (N=199)
Anorexia (Psychiatric disorders) | 1 (1)
General Weakness (General disorders) | 1 (1)
Stroke (Vascular disorders) | 1 (1)
Ankle Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Malignancy Of Unknown Origin (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil (N=199)
Weakness (General disorders) | 3
Anorexia (Psychiatric disorders) | 7
Abdominal Discomfort (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 5
Dizziness (Nervous system disorders) | 7
Headache (Nervous system disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No